CLINICAL TRIAL: NCT04766918
Title: The Effect of Different Molecular Weight of Hyaluronic Acid for Patients With Carpal Tunnel Syndrome
Brief Title: The Effect of Different Molecular Weight of HA for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician and associated professor of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Different molecular HA for CTS
Record Dates: First submitted 2021-02-20; First posted 2021-02-23 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydrodissection; hyaluronic acid
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High molecular weight hyaluronic acid (Experimental): Ultrasound-guided hydrodissection with high molecular weight hyaluronic acid between carpal tunnel and median nerve (total 2 times with one-week interval)
  Interventions: Procedure: Sono-guided injection with high molecular weight hyaluronic acid
- Low molecular weight hyaluronic acid (Active Comparator): Ultrasound-guided hydrodissection with low molecular weight hyaluronic acid between carpal tunnel and median nerve (total 2 times with one-week interval)
  Interventions: Procedure: Sono-guided injection with low molecular weight hyaluronic acid

INTERVENTIONS:
Procedure: Sono-guided injection with high molecular weight hyaluronic acid — Sono-guided injection with hyaluronic acid (Aragan Plus, 20 mg/2 ml, 3000kDa) between carpal tunnel and median nerve
  Arms: High molecular weight hyaluronic acid
Procedure: Sono-guided injection with low molecular weight hyaluronic acid — Sono-guided injection with hyaluronic acid (ARTZDispo, 25 mg/2 ml, 600-1200kDa) between carpal tunnel and median nerve
  Arms: Low molecular weight hyaluronic acid

SUMMARY:
Recently, nerve hydrodissection is utilized to assist ultrasound-guided nerve injection and studies recommend its clinical benefit for peripheral entrapment neuropathy. Hyaluronic acid (HA) can decrease the post-surgery adhesion of soft tissue and nerve but its clinical application in clinical practice is very rare.

We just proved that single HA injection have short-term effectiveness in mild-to-moderate carpal tunnel (CTS) cases and this finding may hint the therapeutic effectiveness of nerve hydrodissection for CTS depend on absorption time of solution. In addition, no study compare different weight of HA for nerve injection so far. Hence, the purpose of this study aim to compare different weight of HA for CTS and whether hydrodissection effect depend on the absorption time of solution or not.

DETAILED DESCRIPTION:
Participants established with diagnosis of mild-to-moderate CTS will been randomly assigned to high molecular weight HA (Aragan Plus, 20 mg/2 ml, 3000kDa) or low molecular weight HA (ARTZDispo, 25 mg/2.5 ml, 600-1200kDa) groups. With ultrasound guidance, total two-sessions of high or low molecular weight HA with one week interval will been injected into intra-carpal region. The Boston Carpal Tunnel Syndrome Questionnaire is assigned as primary outcome. The secondary outcomes encompass visual analog scale, electrophysiological studies, cross-sectional area of the median nerve, mobility of median nerve and absorption time of HA. The assessment is performed prior injection and at 2 week, 1, 2, 3 and 6 months post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 3rd, 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 3rd, 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 3rd, 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of conduction velocity, amplitude of median nerve on 2nd week, 1st, 3rd, 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month
  electrophysiological study of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of mobility of median nerve on 2nd week, 1st, 3rd, 6th month after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month
  Using the musculoskeletal sonogram to measure the mobility of the median nerve before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, School of Medicine, National Defense Medical Center, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Ozgenel GY. Effects of hyaluronic acid on peripheral nerve scarring and regeneration in rats. Microsurgery. 2003;23(6):575-81. doi: 10.1002/micr.10209. PMID 14705074
- [Background] Burns JW, Skinner K, Colt J, Sheidlin A, Bronson R, Yaacobi Y, Goldberg EP. Prevention of tissue injury and postsurgical adhesions by precoating tissues with hyaluronic acid solutions. J Surg Res. 1995 Dec;59(6):644-52. doi: 10.1006/jsre.1995.1218. PMID 8538160
- [Background] Ozgenel GY, Filiz G. Effects of human amniotic fluid on peripheral nerve scarring and regeneration in rats. J Neurosurg. 2003 Feb;98(2):371-7. doi: 10.3171/jns.2003.98.2.0371. PMID 12593625
- [Background] Atzei A, Calcagni M, Breda B, Fasolo G, Pajardi G, Cugola L. Clinical evaluation of a hyaluronan-based gel following microsurgical reconstruction of peripheral nerves of the hand. Microsurgery. 2007;27(1):2-7. doi: 10.1002/micr.20299. PMID 17205576